CLINICAL TRIAL: NCT07331571
Title: Effects of Myofascial Release With and Without Autogenic Inhibition Muscle Energy Technique in Patients With Non-specific Chronic Neck Pain
Brief Title: Myofascial Release With and Without Autogenic Inhibition Muscle Energy Technique in Non-specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0178
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Non Specific Chronic Neck Pain
Keywords: Neck Ache; Myofascial Release Therapy; Autogenic Inhibition Technique; Muscle Energy Technique; Chronic Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release with Autogenic Inhibition Muscle Energy Technique (Experimental)
  Interventions: Other: Autogenic Inhibition Muscle Energy Technique; Other: Myofasical Release Therapy; Other: Standardized Physiotherapy Treatment
- Myofascial Release Therapy (Active Comparator)
  Interventions: Other: Myofasical Release Therapy; Other: Standardized Physiotherapy Treatment

INTERVENTIONS:
Other: Autogenic Inhibition Muscle Energy Technique — AI MET was applied for upper trapezius 5 times for each side, similarly for levator scapulae it was applied 5 times for each side. AI MET was applied for posterior, middle and anterior fibres of scalene muscle. For sternocleidomastoid muscle it was applied for at least twice for each side. 8 sessions were conducted for 6 weeks, with 3 sessions scheduled every week.
  Arms: Myofascial Release with Autogenic Inhibition Muscle Energy Technique
Other: Myofasical Release Therapy — MFR for upper trapezius and levator scapulae was carried out 5 times for each side. A total of 18 sessions were conducted for 6 weeks, with 3 sessions scheduled every week.
Other: Standardized Physiotherapy Treatment — Electric hot pack for 10 minutes for 10 minutes, TENS with frequency of 120Hz at low intensity having pulse duration of 50-200μs for 10 minutes & Grade I and II Maitland posteroanterior central glide with 3 sets of 30 oscillations, for alleviation of pain at the target vertebral segment.

SUMMARY:
The study was conducted to determine the effects of myofascial release therapy with and without autogenic inhibition muscle energy technique in patients with non-specific chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain for at least 3 months
* Pain intensity on NPRS between 4 to 7
* Limited neck range of motion
* Use of computer for at least 2 hours daily
* Negative Sharp-Purser and alar ligaments test (to rule out atlantoaxial instability, integrity of transverse and alar ligaments)

Exclusion Criteria:

* History of trauma
* Cervical spine fracture
* Open neck surgery
* Cervical radiculopathy
* Paresthesia
* Cervical myelopathy
* Rheumatoid Arthritis
* Ankylosing Spondylitis
* Multiple Sclerosis
* Fibromyalgia
* Hemorrhage tendency and/or anticoagulation treatment
* Whiplash Injury

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment to the end of treatment at 6 weeks
  Numeric Pain Rating Scale is utilized to evaluate pain. It consists of 11 points, having an overall score ranging from 0 and 10, where: 0 represents no pain, 1 - 3 represents mild pain, 4 - 6 represents moderate pain and 7 - 10 represents the most severe pain.
Neck Disability Index | From enrollment to the end of treatment at 6 weeks
  Neck Disability Index is a questionnaire that has 10-questions for determining cervical pain and functional disability linked with the activities of daily living. It consists of questions on pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Scores in each item is described in 6 stages, from 0 to 5 points. The total of 0-4 points indicate no disability, 5-14 points indicate mild disability, 15-24 points indicate moderate disability, 25-34 points indicate severe disability and 35-50 points indicate complete disability

SECONDARY OUTCOMES:
ROM Cervical Spine (Flexion) | From enrollment to the end of treatment at 6 weeks
  Changes in cervical spine flexion ROM at baseline and 6th week of intervention was measured using goniometer.
ROM Cervical Spine (Extension) | From enrollment to the end of treatment at 6 weeks
  Changes in cervical spine extension ROM at baseline and 6th week of intervention was measured using goniometer.
ROM Cervical Spine (Lateral Flexion) Left Side | From enrollment to the end of treatment at 6 weeks
  Changes in cervical spine lateral flexion on left side ROM at baseline and 6th week of intervention was measured using goniometer.
ROM Cervical Spine (Lateral Flexion) Right Side | From enrollment to the end of treatment at 6 weeks
  Changes in cervical spine lateral flexion on right side ROM at baseline and 6th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Left Side | From enrollment to the end of treatment at 6 weeks
  Changes in cervical spine rotation on left side ROM at baseline and 6th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Right | From enrollment to the end of treatment at 6 weeks
  Changes in cervical spine rotation on right side ROM at baseline and 6th week of intervention was measured using goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Shakil ur Rehman, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- Rehab Max Physio & Sports Injury Clinic, Layyah, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No